CLINICAL TRIAL: NCT01332864
Title: Physiological and Behavioral Effects of Osteopathic Manipulative Treatment on Patients With Chronic Headache: A Randomized Clinical Trial
Brief Title: Effect of Osteopathic Manipulative Treatment for Patients With Chronic Headache
Acronym: OMTHA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Responsible Party: Principal Investigator, Michael Seffinger, Principal Investigator, Associate Professor and Chair of Dept. of NMM/OMM, Western University of Health Sciences
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CV4OMTHA
Record Dates: First submitted 2011-04-04; First posted 2011-04-11 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Headache; Cephalgia; Migraine
Keywords: headache; migraine; cephalgia; osteopathic manipulative treatment
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Manipulation, Osteopathic; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- OMT to the head and rest of body (Active Comparator): OMT is the intervention that will be applied to areas of somatic dysfunction as well as to the head using a compression of the fourth ventricle (CV4) technique.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)
- Light touch (Placebo Comparator): Light touch will be applied to the head region for 10 minutes with the patient at rest in the supine position.
  Interventions: Procedure: Light touch
- OMT with CV4 to head (Experimental): OMT is the intervention using the CV4 technique to the head region for 10 minutes with patient at rest.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)
- OMT to the body except the head region (Active Comparator): OMT is the intervention that will be applied to areas of somatic dysfunction in any region except the head.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment (OMT) — O OMT applied to areas of somatic dysfunction other than the head region.
  Other Names: headache; OMT; somatic dysfunction ICD-9 code 739.0
  Arms: OMT to the body except the head region; OMT to the head and rest of body; OMT with CV4 to head
Procedure: Light touch — Light touch applied to head region for 10 minutes with patient supine at rest.
  Other Names: placebo; sham
  Arms: Light touch

SUMMARY:
Participants with chronic or recurrent headache, unrelated to any known pathology or disease, will be randomly assigned to one of four interventions: Osteopathic manipulation of the body other than the head, osteopathic manipulation of the head, osteopathic manipulation of the head and rest of the body, or light touch on the head only but no manipulation. Measurements of heart rate and blood pressure variability, peripheral blood flow, and behavioral changes, such as mood, pain duration, intensity and frequency will be assessed.

DETAILED DESCRIPTION:
Sixty subjects will be recruited to participate in the study via word of mouth and mass email notification of employees and students at Western University of Health Sciences in Pomona, CA.

Patients will be randomly assigned to 1 of 4 groups for a specific Osteopathic Manipulative Treatment (OMT): Compression of Fourth Ventricle (CV4) only, CV4 and subject appropriate OMT, subject appropriate OMT only (no CV4), and sham (touch only). There will be 8 subjects per OMT group, making it 24 subjects altogether assigned to one of the three OMT groups, and 24 sham subjects.

Power analysis for determination of sample sizes: The investigators have no data on preliminary studies of the effect of OMT on chronic headaches, and there is only one study of the immediate effect on tension type headache patients after CV4, so power analysis is a rough estimate at this point for the one week headache symptom evaluation post OMT. From preliminary studies in this lab, the investigators can expect for 'CV4 only' 80% of participants to have significant still point objective response vs sham treatment which the investigators expect will significantly effect about 10% of the participants. There needs to be at least 16 subjects in each of two groups assessing this outcome measure, so 16 receiving CV4 and 16 sham to detect the 70% difference in still point measure. To detect differences between any OMT and sham, since there are three groups receiving OMT of some type, when the investigators consider how many in each of these three groups vs the sham group, the investigators figured 8 per each OMT group, of which 2 are CV4 (thus 16 get CV4), making it 24 subjects in the combined OMT groups. Therefore, the investigators need 24 sham subjects to make it equal numbers for balanced analysis (OMT vs sham), and to detect differences in the OMT interventions and sham interventions. Considering a possibility of 25%, or 12 subjects, not responding to the follow up survey at one week, the investigators figured recruitment of 60 subjects would ensure the investigators would have enough to make our calculations and be able to determine if there are significant differences between groups.

The investigators have no preliminary studies on the effect of OMT or sham on mood in patient with headaches, so this part of the study is an exploratory assessment and sample size calculations will be able to be performed with the data gathered from this study for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* chronic or recurrent headaches at least as often as one time per week

Exclusion Criteria:

* recent head trauma
* brain disease or pathology
* seizure disorder
* using beta or alpha blocker medications
* allergy to sticky tape used to affix leads to skin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Head pain frequency | one week after intervention
  seven days after the intervention participants will be called by telephone and asked whether they had their usual headache in the week following the intervention.

SECONDARY OUTCOMES:
Head pain intensity | one week
  one week after intervention participants will be contacted and asked to rate the intensity of their headaches after the intervention.
Head pain duration | one week
  one week after the intervention participants will be contacted and asked the duration of the headaches.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Seffinger, D.O., Principal Investigator — Western University of Health Sciences
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

REFERENCES:
- See also: Western University web site — http://www.westernu.edu